CLINICAL TRIAL: NCT06062056
Title: Leveraging Community-based Behavioral Health to Increase Vaccine Uptake in Latinx Adults With Mental Illness
Brief Title: Motivational Interviewing for Vaccine Uptake in Latinx Adults
Acronym: MIVacuna
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: It's focus on vaccine hesitancy did not align with the administration's philosophy
Sponsor: Boston College (Other)
Collaborators: East Boston Neighborhood Health Center (Unknown); Harvard School of Public Health (HSPH) (Other); Boston Children's Hospital (Other); National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Health Services Research
Other Study IDs: 23.049.01; 5R01NR020482 (NIH)
Record Dates: First submitted 2023-08-03; First posted 2023-10-02 (Actual); Last update posted 2025-09-15 (Actual); Status verified 2025-09

CONDITIONS: Vaccine Hesitancy
Keywords: COVID-19; Influenza; Latinx; Behavioral health; Motivational interviewing
MeSH Terms: conditions — Vaccination Hesitancy; COVID-19; Influenza, Human | interventions — Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: A pragmatic multiple-period, cluster-randomized crossover design will be used.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Behavioral health clinicians will use motivational interviewing with eligible patients to address vaccine hesitancy
  Interventions: Other: EHR alert; Behavioral: Motivational Interviewing; Behavioral: Warm hand off to nurse
- Control (No Intervention): Control sites will adhere to standard practice in behavioral health sessions (i.e., no discussions about vaccination)

INTERVENTIONS:
Other: EHR alert — An EHR alert will be fired if a behavioral health patient is missing a COVID-19 or influenza vaccine.
  Arms: Intervention
Behavioral: Motivational Interviewing — In response to the alert and using support tools in the EHR, the behavioral health clinician will integrate motivational interviewing into the counseling session to discuss vaccine hesitancy (if it is deemed appropriate based on patient needs and clinical judgment).
  Arms: Intervention
Behavioral: Warm hand off to nurse — For patients interested in vaccination following motivational interviewing, the behavioral health clinician will do a warm hand off to a nurse for vaccination
  Arms: Intervention

SUMMARY:
The goal of this clinical trial is to test whether modified behavioral health services, integrating motivational interviewing, will reduce vaccine hesitancy and increase uptake for the COVID-19 and influenza vaccines among Latinx adults with mental illness.

DETAILED DESCRIPTION:
Prior to the Coronavirus disease (COVID-19) pandemic, the World Health Organization declared vaccine hesitancy, defined as a delay in the acceptance or refusal of vaccination despite availability of vaccination services, as one of the top 10 threats to global health. Today, despite massive recent and ongoing global efforts, vaccine hesitancy remains a major threat, particularly in populations that experience health disparities rooted in structural racism. One such population is Hispanic/Latinx adults (Latinxs). Prior to the national COVID-19 vaccine campaign, Latinxs had twice the rate of COVID-19 infection, 2.8 times the rate of hospitalization and 2.3 times the death rate of non-Latinx whites. Despite being at higher risk of COVID-19 related morbidity and mortality, Latinxs have been particularly hesitant to get vaccinated. In the early stages of vaccine rollout, vaccine uptake rates among Latinxs lagged at least 10% percentage points behind non-Latinxs and, as of Feb 2022, only 37% of Latinxs compared to 56% of non-Latinx whites had received a booster shot.

Adults with mental illness are also at high risk for COVID-19 infection, with more severe complications and higher mortality Yet there are no strategies for addressing vaccine hesitancy in this population. This gap is particularly important for Latinxs, who have disproportionately borne the mental health burden of the pandemic. There is, therefore, an urgent need for innovative, practical, and sustainable strategies to address vaccine hesitancy among the priority population of Latinx adults with mental illness.

The investigators will address this gap with a novel intervention that integrates evidence-based motivational interviewing (MI) into behavioral health (BH) services, coupled with electronic prompting, and vaccination access at the point of care. Key to the intervention is that the proposed MI protocol explicitly acknowledges cultural values that are central to the Latinx population and impact their interactions with health care providers. Additionally, the intervention has been specifically designed to: (i) be feasible and readily implemented in an integrated care setting, such as that offered by federally qualified health centers (FQHC); (ii) be sustainable in the long-term regardless of how the rapidly-changing COVID-19 vaccination landscape evolves; and, (iii) provide additional potential benefits in the form of increasing influenza vaccination which is generally low in the Latinx population.

ELIGIBILITY:
Patient Inclusion Criteria:

* Aged 18 years and older
* Identifies as Latinx or speaks Spanish
* Completed an eligible behavioral health (BH) visit between the start and end dates of the intervention period.
* Patient is missing a COVID-19 vaccine/booster or the influenza vaccine at the beginning of their behavioral health visit (i.e., they are not fully up to date with their COVID-19 and influenza vaccines)

Patient Exclusion Criteria:

- NA

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 3698 (Actual)
Dates: Start 2023-10-02 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Received COVID-19 vaccine/booster following an eligible behavioral health visit | Within 6 weeks of an eligible behavioral health visit
  Binary indicator extracted from EHR
Received influenza vaccine following an eligible behavioral health visit | Within 6 weeks of an eligible behavioral health visit
  Binary indicator extracted from EHR

SECONDARY OUTCOMES:
Survey measure of vaccine hesitancy | Completed within one week of an eligible behavioral health visit
  Survey items measuring the 3Cs (complacency, confidence, convenience) of vaccine hesitancy
Survey measure of provider trust | Completed within one week of an eligible behavioral health visit
  Survey item assessing if patients trust that their counselor will give them accurate vaccine (COVID-19 or influenza) information. Developed by research team.
Survey measure of vaccination intention | Completed within one week of an eligible behavioral health visit
  Survey items assessing whether patient intends to get a vaccine (COVID-19 or influenza). Developed by the research team.

OTHER OUTCOMES:
COVID-19 vaccine series initiation (at least one dose of the vaccine) | 12 month intervals over a total of 48 months
  Binary indicator extracted from EHR assessed longitudinally
Up to date with COVID-19 vaccination (consistent with CDC guidelines) | 12 month intervals over a total of 48 months
  Binary indicator extracted from EHR assessed longitudinally
Up to date with influenza vaccine; received vaccine for current season (consistent with CDC guidelines) | 12 month intervals over a total of 48 months
  Binary indicator extracted from EHR assessed longitudinally

CONTACTS AND LOCATIONS:
Overall Officials: Kirsten Davison, PhD, Principal Investigator — Boston College
Locations (2):
- United States (2):
  - South End Community Health Center, Boston, Massachusetts
  - East Boston Neighborhood Health Center, Boston, Massachusetts

IPD SHARING:
Plan to Share IPD: No
We submitted our application for review prior to the implementation of the new data sharing guidelines (January 25, 2023)

REFERENCES:
- [Background] Scrivano RM, van de Water BJ, Rueras N, Alfonso J, McManama O'Brien KH, Soto X, Caumeran VJS, Campos BM, Mancusi M, Diehl B, Southwick E, Moreno E, Bora C, Armbruster S, Abuelezam NN, Calvo R, Haneuse S, Davison KK. Motivational Interviewing for Vaccine Uptake in Latinx Adults (MI Vacuna): Study protocol for a pragmatic multiple-period cluster-randomized crossover trial. Contemp Clin Trials. 2025 Aug;155:107987. doi: 10.1016/j.cct.2025.107987. Epub 2025 Jun 14. PMID 40523466
- See also: Research team website — https://www.bc.edu/content/bc-web/schools/ssw/sites/labs/thrive-lab/mi-vacuna.html